CLINICAL TRIAL: NCT02256228
Title: Peroperative Analgesia Following Cytoreductive Surgery. A Randomized, Double-blind, Comparison Between Intra-peritoneal Local Anesthesia and Placebo - Multicenter Study
Brief Title: Intra-Peritoneal Local Anaesthesia After Cytoreductive Surgery
Acronym: IPLA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IPLA-CRS
Record Dates: First submitted 2014-10-01; First posted 2014-10-03 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Pain
Keywords: Analgesia; Local infiltration analgesia; Pain, relief; Pain, Postoperative; Intra-peritoneal analgesia; Ropivacaine; Saline; Therapeutic Uses; Analgesics, Non-Narcotic; Analgesics; Opioids; Morphine; Pain; Postoperative Complications; Physiological Effects of Drugs; Anesthetics, Local; Anesthetic; Cytoreductive; Surgery; Cancer
MeSH Terms: conditions — Pain; Agnosia; Pain, Postoperative; Postoperative Complications; Neoplasms | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group R (Active Comparator): Ropivacaine is instillated through one multi-hole catheter wich would be inserted percutaneously in all patients and tunnelled about 1-2 cm lateral to the abdominal incision and the tip of the catheter placed in the intra-peritoneal cavity. The catheter would not be ligated and fixed in situ intra-peritoneally. Twenty ml of Ropivacaine would be injected subcutaneously along both sides of the incision prior to skin closure. Additionally, 20 ml of Ropivacaine (1mg/mL) would be injected every hour by an automatic pump via the intra-peritoneal catheter into the abdomen.
  Interventions: Drug: Ropivacaine
- Group P (Placebo Comparator): Saline is instillated through one multi-hole catheter wich would be inserted percutaneously in all patients and tunnelled about 1-2 cm lateral to the abdominal incision and the tip of the catheter placed in the intra-peritoneal cavity. The catheter would not be ligated and fixed in situ intra-peritoneally. Twenty ml of Saline would be injected subcutaneously along both sides of the incision prior to skin closure. Additionally, 20 ml of Saline would be injected every hour by an automatic pump via the intra-peritoneal catheter into the abdomen.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Ropivacaine — Active Group
  Other Names: Narop
  Arms: Group R
Drug: Saline — Placebo Comparator
  Other Names: Sodium Chloride
  Arms: Group P

SUMMARY:
Can perioperative administration of intra-peritoneal local anaesthetics further reduce postoperative pain, inflammation and outcome in patients undergoing major abdominal surgery (cytoreductive surgery) and managed with thoracic epidural analgesia? - Multicenter study.

DETAILED DESCRIPTION:
The aim of this study is to measure the efficacy of local anesthetics (LA) administered into the intra-peritoneal cavity compared to placebo. Our hypothesis is that the injection of local LAs intra-peritoneally would reduce post-operative pain and the inflammatory process caused by the massive release of cytokines during extensive cytoreductive surgery. The study is a controlled, parallel group, double blind, prospective, randomized and performed at Sahlgrenska University Hospital in Goteborg, Sweden . Twenty mL of ropivacaine or saline would be injected every hour by an automatic pump via the intra-peritoneal catheter into the abdomen according to group randomization in order to double blind patients and all personnel involved in the study.

The parameters that would be evaluated are inflammatory markers, postoperative morbidity, pain intensity, consumption of morphine, cognitive function and progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

- Patients with widespread malignant intra-abdominal ovary cancer stadium III-IV and are operated by extensive resection of intra-abdominal viscera as well as the parietal peritoneum (cytoreductive surgery, CRS)

Exclusion Criteria:

* Body mass index > 35
* American Society of Anesthesiologists classification > 3
* Renal dysfunction
* Allergic to acetylsalicylic acid
* Unwilling to provide informed consent

Ages: 18 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-10; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Inflammatory Markers | 0-48 hours postoperatively
  Analysis of the following inflammatory markers with Multiplex: IL(interleukin)-1β, IL-1rα, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-9, IL-10, IL-12 (p70), IL-13, IL-15, IL-17A, zBasic FGF (Fibroblast Growth Factor), Eotaxin, G-CSF (granulocyte colony stimulating factor), GM-CSF granulocyte macrophage colony stimulating factor), IFN-γ (interferon), IP-10 (immune protein), MCP-1 (monocyte chemotactic protein), MCAF (monocyte chemotactic and activating factor), MIP-1α (macrophage inflammatory protein), MIP-1β, PDGF-BB (platelet-derived growth factor), RANTES (regulated on activation, normal T cell expressed and secreted), TNF-α (tumor necrosis factor), VEGF (vascular endothelial growth factor)

SECONDARY OUTCOMES:
Postoperative Morphine consumption | 0-48 hours postoperatively
  Total amount of Morphine consumed during the first 48 hours after surgery
Pain Intensity | 0-48 hours postoperatively
  Pain Intensity is measured with Numeric Rating Score 0-10
Cognitive Function | 0-1 month postoperatively
  Patients will complete the following neurophysiological tests upon entering the study and within one month after surgery: Verbal Learning Test (VLT), Concept Shifting Test (CST), Letter-Digit Coding, Verbal Learning Test - Delayed Recall (VLT-D)
Progression-free Survival | 0-3 years postoperatively
  Progression-free Survival measures the length of time after treatment during which the cancer being treated does not get worse.
Postoperative Morbidity/Complications | 0-30 days postoperatively
  Measuring the numbers of Postoperative Morbidity/Complications within one month after surgery:
  Morbidity:
  * Local infections
  * Urinary infection (urine culture)
  * Pneumonia (X-ray, C-reactive protein, Fever)
  * Sepsis (Fever, Leucocyte count in blood, Heart Rate, Respiratory Rate)
  * Pleural fluid (X-ray verified)
  * Deep Vein Thrombosis (D-dimer, ultrasound verified)
  * Pulmonary embolism (Computed Tomography/ Scint-X)
  * Acute Myocardial Infarction (Electrocardiography, Troponin I)
  * Atrial fibrillation or serious arrhythmia during the first 48 hours after surgery (Electrocardiography)
  * Respiratory failure (prolonged mechanical ventilation)
  * Renal failure (Serum Creatinine, Diuresis, AKIN criteria)
  * Inotropic needs > 12 hours after surgery
  Surgical Complications:
  * Intraabdominal bleeding
  * Leakage from anastomosis
  * Abdominal abscess
  * Paralytic ileus
  * Pancreatic leakage (requiring drainage)

CONTACTS AND LOCATIONS:
Overall Officials: Sven-Egron Thorn, MD PhD, Principal Investigator — Dept. of Anesthesia and Intensive Care, Sahlgrenska University Hospital, Goteborg, Sweden; Anil Gupta, MD PhD, Study Chair — Dept. of Anesthesia and Intensive Care, Orebro University Hospital, Orebro, Sweden; Sven-Erik Ricksten, MD PhD, Study Chair — Dept. of Anesthesia and Intensive Care, Sahlgrenska University Hospital, Goteborg, Sweden
Locations (1):
- Dept. of Gynecological Surgery and Anesthesia and Intensive Care, Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Derived] Hayden JM, Oras J, Block L, Thorn SE, Palmqvist C, Salehi S, Nordstrom JL, Gupta A. Intraperitoneal ropivacaine reduces time interval to initiation of chemotherapy after surgery for advanced ovarian cancer: randomised controlled double-blind pilot study. Br J Anaesth. 2020 May;124(5):562-570. doi: 10.1016/j.bja.2020.01.026. Epub 2020 Mar 13. PMID 32172954
- [Derived] Hayden J, Gupta A, Thorn SE, Thulin P, Block L, Oras J. Does intraperitoneal ropivacaine reduce postoperative inflammation? A prospective, double-blind, placebo-controlled pilot study. Acta Anaesthesiol Scand. 2019 Sep;63(8):1048-1054. doi: 10.1111/aas.13410. Epub 2019 Jun 17. PMID 31206591